CLINICAL TRIAL: NCT05008718
Title: Silver Diamine Fluoride: A Randomized Controlled Trial on Its Effectiveness As A Caries Arresting Agent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Intan Elliayana Binti Mohammed, Principal Investigator, Dr, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDF_UiTM
Record Dates: First submitted 2021-08-14; First posted 2021-08-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dental Caries; Quality of Life
Keywords: silver diamine fluoride; dental caries; effectiveness
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 38% SDF group (Active Comparator): 38% silver diamine fluoride will be applied on caries lesions on deciduous teeth with a minimum score of 05 as defined by the International Caries Detection and Assessment System (ICDAS)
  Interventions: Other: 38% SDF group
- 5% NaF group (Placebo Comparator): 5% sodium fluoride will be applied on caries lesions on deciduous teeth with a minimum score of 05 as defined by the International Caries Detection and Assessment System (ICDAS)
  Interventions: Other: 5% NaF group

INTERVENTIONS:
Other: 38% SDF group — Participants will be randomized and will receive either 38% SDF treatment or 5% NaF treatment
  Arms: 38% SDF group
Other: 5% NaF group — Participants will be randomized and will receive either 38% SDF treatment or 5% NaF treatment
  Arms: 5% NaF group

SUMMARY:
The aim of the study is to assess the effectiveness of 38% Silver Diamine Fluoride (SDF) solution and to determine if it is superior to 5% NaF varnish in arresting carious lesions in the primary teeth of young children attending general dental clinic, Universiti Teknologi Mara.

Hypothesis: Topical application of a 38% SDF solution on the primary teeth is superior to that of a 5% NaF varnish in arresting caries lesions in children at 3-months follow-up

An intervention study is planned to compare the effectiveness of 38% SDF and 5% NaF in arresting caries lesions in primary teeth of 3-8 years old children attending general dental clinic, Universiti Teknologi Mara. The sample size needed (considering a 20% dropout rate) is 66 participants in each group. In addition, this study also aims to determine the demographic background, oral health-related habits, oral health-related quality of life of the participants and the parents acceptance on SDF treatment towards their child.

DETAILED DESCRIPTION:
Convenience sampling will be used, in which patient will be recruited from General Dental Clinic (Sapphire), Faculty of Dentistry, Universiti Teknologi Mara. The total number of participants needed is 132. At baseline, during the screening and examination stage, apart from ICDAS score and the decayed, missing, and filled surface (dmfs) index to record each child's caries experience, recorded status will also include baseline bitewings of posterior teeth and DIAGNOdent reading (triplicate reading will be carried out to achieve accurate value) for all lesions. Periapical radiograph of anterior teeth will only be taken to confirm no pulp involvement when depth of lesion is questionable. Five tooth surfaces (buccal, lingual, mesial, distal and occlusal) will be examined in each posterior tooth and four tooth surfaces (labial, lingual, mesial and distal) in each anterior tooth. A carious lesion will be recorded as active if softness is detected upon gentle probing. If the lesion is hard when probing, it will be classified as an arrested caries. Screening and oral examination will be conducted on a dental chair in assigned clinic at Faculty of Dentistry, Universiti Teknologi Mara, primarily through careful visual inspection with the aid of a World Health Organization (WHO) CPI probe and a stainless steel/disposable front surface dental mirror by the main researcher. The main researcher will record each patient's caries status on a separate paper-based trial record at the beginning of the study in which she will not have the access to Integrated Dental Record Management System (IDERMS) in order to maintain blindness. Before conducting the study, a training and calibration session for oral examination (ICDAS and DIAGnodent utilization) is planned for the main researcher with one specialist in dental public health and one specialist in paediatric dentistry with the aim to achieve the kappa values of inter and intra-reliability ≥0.8.

Next, after the screening and before consent, if the child is eligible for the study, parents or guardians will be provided with information about SDF and NaF, follow-up instructions, oral hygiene instruction and diet education which will use video and pamphlet. Parents and guardians who agreed to participate in the study will be given questionnaire which include children's demographic background, oral-health related habits, and Malay- ECOHIS together with the information sheet and consent sheet. Appointment for first topical fluoride application will be given within one week from baseline oral examination day.

On the first appointment day, the allocation of patient between 38% SDF application and 5 % NaF application is randomized using sequentially numbered, opaque sealed envelopes (SNOSE) procedure (Doig & Simpson, 2005). Block of four and six will be used to ensure that similar numbers of patients are enrolled into each group and to ensure the prediction of allocation sequence impossible. The order of the blocks will be determined by flipping a coin. This will be carried out by a dental officer/postgraduate student who is not involved with the study. He/she will keep the piles of blocks and when participant comes for the intervention, he/she will ask the operator to select one envelope from the first pile of blocks according to allocated sequence and will prepare the treatment selected. After first application is completed, he/she also will be the one who will update the Integrated Dental Record Management System (IDERMS) on which treatment has been used for the respective participants in order for him/her to prepare the same treatment for the 1-month follow up. The topical fluoride applications will be carried out by the other three researchers who are not involved in the screening and assessing of the lesion activity. Before the study, they will be trained by a paediatric dental specialist who is not involved in the study for the clinical application procedure. This is a double-blind clinical trial where the main researcher is not aware of which treatment the participants will be receiving, the other researchers are not aware which treatment they are providing and participants are not aware of which treatment they are receiving.

Participants will be called again for second application of same treatment they received on the first appointment after one month. Final appointment follow-up examination will be given at three months after first application of the topical fluoride. Same examiner will conduct the follow-up oral examinations using the same equipment, procedure and diagnostic criteria as those used in the baseline examination. Another questionnaire inclusive of parental acceptability for SDF treatment on their children and OHRQoL (Malay-ECOHIS) will be distributed to the same parents or guardians and will be asked to complete the questionnaire survey. After study is completed, the participants will be assigned back to undergraduate students for definitive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Three to eight years old children. The reason for selecting children up to eight years old is because there are still patients aged seven to eight years old who presented with posterior deciduous teeth and upper lateral incisor deciduous teeth caries. Children below three years old are not included in order to obtain better cooperation from the participants.
* Children who are generally healthy, not medically compromised
* Children who have at least one active carious lesion on a deciduous tooth which include upper anterior teeth caries (c-c) with a minimum score of 05 as defined by the International Caries Detection and Assessment System (ICDAS)
* Provision of informed consent by the parent or guardian

Exclusion Criteria:

* Children with spontaneous or elicited pain from caries, tooth mobility, or signs of pulpal infection
* Children with severe medical conditions that would not allow management in the clinic
* Children with hereditary developmental defects, such as amelogenesis imperfecta
* Children with known allergies or sensitivities to dental materials, including silver diamine fluoride and sodium fluoride
* Inability to cooperate for silver diamine fluoride treatment or return for recall visits 3 months

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Caries arrest rate | 3 months
  After SDF or NaF application, after 3 months assessment, smooth and hard tooth surface that could not be penetrated by probe easily will be classified as arrested lesion. Caries arrest rate will be calculated by the percentage of all arrested lesions over all treatment applied teeth in respective arm.
  DIAGNOdent reading will be taken for all lesions before and after treatment in which DIAGNOdent reading ≥ 16 is indicated more likely to develop dentin caries after 24 mos.

SECONDARY OUTCOMES:
Oral Health-Related Quality of Life | 3 months
  Participants' oral health-related quality of life will be assessed using ECOHIS (Early Childhood Oral Health Impact Scale) that has been translated and validated in Malay language. Parents will be given the questionnaire and will be asked to complete it before and after intervention.
  The Malay-ECOHIS consists of 13 items with two main parts: the child impacts section (CIS) which has 4 domains with 9 items and the family impacts section (FIS) which has 2 domains with 4 items. The total of Malay-ECOHIS scores and scores for individual domains will be calculated as a simple sum of the response codes. Higher scores will indicate greater degrees of oral impact on the quality of life of the child.

OTHER OUTCOMES:
Parental acceptance on SDF treatment | 3 months
  Parents will be given questionnaire regarding their acceptance on SDF treatment being applied at their children after intervention is completed at 3 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Intan Elliayana binti Mohammed, Principal Investigator — Faculty of Dentistry, Universiti Teknologi Mara
Locations (1):
- Faculty of Dentistry, Universiti Teknologi Mara, Sg. Buloh Campus, Sungai Buloh, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No